CLINICAL TRIAL: NCT02348177
Title: A Pharmacokinetics Study Comparing Lopinavir Plasma Exposure When Given as Lopinavir/Ritonavir (1:1) in the Presence of Rifampicin and Lopinavir/Ritonavir (4:1) Without Rifampicin in HIV and TB Co-infected Children in South Africa.
Brief Title: Pharmacokinetics of Lopinavir/Ritonavir Superboosting in Infants and Young Children Co-infected With HIV and TB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: University of Cape Town (Other); Medecins Sans Frontieres, Netherlands (Other); French Development Agency (Other Government); UBS Optimus Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDiHIVPed001
Record Dates: First submitted 2014-12-03; First posted 2015-01-28 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Acquired Immunodeficiency Syndrome; Tuberculosis
Keywords: Human immunideficiency virus; Tuberculosis; superboosting; lopinavir/ritonavir 1:1; Pediatric TB/HIV co-infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TB/HIV co-infection (Experimental): Superboosting lopinavir with ritonavir in 1:1 ratio during TB/HIV co-infection and treatment of HIV with lopinavir/ritonavir 4:1
  Interventions: Drug: lopinavir with ritonavir in 1:1 ratio; Drug: Lopinavir/ritonavir 4:1

INTERVENTIONS:
Drug: lopinavir with ritonavir in 1:1 ratio — During co-treatment of rifampicin containing tuberculosis treatment and lopinavir/ritonavir (4:1) based therapy, additional ritonavir is given to make lopinavir/ritonavir 1:1 ratio
  Other Names: Lopinavir/ritonavir; Ritonavir
Drug: Lopinavir/ritonavir 4:1 — This is the conventional dosing of LPV/r 4:1 for HIV when TB treatment has not been started or has been stopped
  Other Names: Lopinavir/ritonavir

SUMMARY:
The purpose of this study is to determine the lopinavir levels in blood of HIV and TB infected children (3-15kg) when given lopinavir/ritonavir in a 1:1 ratio with rifampicin containing TB regimen and its safety.

DETAILED DESCRIPTION:
This is a multicentre, open label, non-randomized, prospective, noninferiority study to compare the pharmacokinetics of lopinavir administered with superboosting (LPV/r 1:1) and concurrent RIF treatment or with standard boosting (LPV/r 4:1) without concurrent RIF treatment, and to assess the safety, tolerance, and virological effect of superboosting in HIV-TB co-infected infants and children weighing >3 kg and ≤15 kg.

LPV/r will be administered as the liquid 80/20 mg/mL formulation (4:1 standard boosting ratio). During anti-TB treatment, additional RTV liquid formulation will be provided to deliver a 1:1 superboosting ratio of LPV to RTV. Actual doses for antiretrovirals and anti-TB drugs will be based on the South African (SA) weight band dosing recommendations and provided as per the site standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of a confirmed diagnosis of HIV-1 infection following SA clinical guidelines
* Weight >3kg ≤15 kg at enrolment
* > 42 weeks gestational age
* On LPV/r-based therapy or about to start a LPV/r-based antiretroviral combination therapy with 2 NRTIs [ABC+3TC or AZT+3TC or d4T+3TC]
* Clinical diagnosis of TB requiring RIF-based therapy
* Parent or legal guardian able and willing to provide written informed consent and able to attend study visits.

Exclusion Criteria:

* For neonates, less than 42 weeks gestation and 14 days old
* Concomitant/chronic treatment with potent enzyme-inducing/inhibiting drugs other than those in the study treatments . See Appendix E (minor inducers/inhibitors and drugs used as part of management of the condition are allowed eg. Steroids)
* Anticipation at the start that anti-TB treatment duration will be longer than 9 months
* Any other condition/finding that, in the investigator's opinion, would compromise the child's participation in this study eg. alanine transferase (ALT) more than 10 times upper limit of normal (ULN), or chronic renal, hepatic or gastrointestinal disease such as malabsorption.
* Children with known malignancies and contraindications to taking LPV/r
* Treatment with experimental drugs for any indication within 30 days prior to study entry; participation in another study may be approved by the study team.

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Modelled C0/morning trough | Predose
  Proportions of children treated with modelled lopinavir morning C0/morning trough <1mg/L at each of the intensive PK evaluations.

SECONDARY OUTCOMES:
C0/morning trough | Predose
  Proportions of children with observed lopinavir morning trough, C0/morning trough <1mg/L at each of the intensive PK evaluations
ALT | baseline, PK1, PK2, PK3
  Safety and tolerability of superboosting focusing on liver functions through clinical and biochemical monitoring.
ECG | baseline, 2 weeks after LPV/r 1:1, PK1
  Potential superboosting cardiac effect monitored by electrocardiogram at the beginning of anti-TB and HIV concomitant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cotton, Professor, Principal Investigator — University of Stellenbosch
Locations (5):
- South Africa (5):
  - The Children's Infectious Disease Clinical Research Unit; University of Stellenbosch, Cape Town, Western Cape
  - Enhancing Care Foundation; Wendworth Hospital, Durban
  - Perinatal HIV Research Unit, Johannesburg
  - Shandukani Research WRHI, Johannesburg
  - Empilweni Services and Research Unit, Johannesburg

REFERENCES:
- [Background] Newell ML, Coovadia H, Cortina-Borja M, Rollins N, Gaillard P, Dabis F; Ghent International AIDS Society (IAS) Working Group on HIV Infection in Women and Children. Mortality of infected and uninfected infants born to HIV-infected mothers in Africa: a pooled analysis. Lancet. 2004 Oct 2-8;364(9441):1236-43. doi: 10.1016/S0140-6736(04)17140-7. PMID 15464184
- [Background] Johnson LF, Davies MA, Moultrie H, Sherman GG, Bland RM, Rehle TM, Dorrington RE, Newell ML. The effect of early initiation of antiretroviral treatment in infants on pediatric AIDS mortality in South Africa: a model-based analysis. Pediatr Infect Dis J. 2012 May;31(5):474-80. doi: 10.1097/INF.0b013e3182456ba2. PMID 22189531
- [Background] Marston M, Becquet R, Zaba B, Moulton LH, Gray G, Coovadia H, Essex M, Ekouevi DK, Jackson D, Coutsoudis A, Kilewo C, Leroy V, Wiktor S, Nduati R, Msellati P, Dabis F, Newell ML, Ghys PD. Net survival of perinatally and postnatally HIV-infected children: a pooled analysis of individual data from sub-Saharan Africa. Int J Epidemiol. 2011 Apr;40(2):385-96. doi: 10.1093/ije/dyq255. Epub 2011 Jan 18. PMID 21247884
- [Background] Gurumurthy P, Ramachandran G, Hemanth Kumar AK, Rajasekaran S, Padmapriyadarsini C, Swaminathan S, Bhagavathy S, Venkatesan P, Sekar L, Mahilmaran A, Ravichandran N, Paramesh P. Decreased bioavailability of rifampin and other antituberculosis drugs in patients with advanced human immunodeficiency virus disease. Antimicrob Agents Chemother. 2004 Nov;48(11):4473-5. doi: 10.1128/AAC.48.11.4473-4475.2004. PMID 15504887
- [Background] McIlleron H, Ren Y, Nuttall J, Fairlie L, Rabie H, Cotton M, Eley B, Meyers T, Smith PJ, Merry C, Maartens G. Lopinavir exposure is insufficient in children given double doses of lopinavir/ritonavir during rifampicin-based treatment for tuberculosis. Antivir Ther. 2011;16(3):417-21. doi: 10.3851/IMP1757. PMID 21555825
- [Background] Zanoni BC, Phungula T, Zanoni HM, France H, Feeney ME. Impact of tuberculosis cotreatment on viral suppression rates among HIV-positive children initiating HAART. AIDS. 2011 Jan 2;25(1):49-55. doi: 10.1097/QAD.0b013e32833f9e04. PMID 20935555
- [Background] Violari A, Cotton MF, Gibb DM, Babiker AG, Steyn J, Madhi SA, Jean-Philippe P, McIntyre JA; CHER Study Team. Early antiretroviral therapy and mortality among HIV-infected infants. N Engl J Med. 2008 Nov 20;359(21):2233-44. doi: 10.1056/NEJMoa0800971. PMID 19020325
- [Background] Reitz C, Coovadia A, Ko S, Meyers T, Strehlau R, Sherman G, Kuhn L, Abrams EJ. Initial response to protease-inhibitor-based antiretroviral therapy among children less than 2 years of age in South Africa: effect of cotreatment for tuberculosis. J Infect Dis. 2010 Apr 15;201(8):1121-31. doi: 10.1086/651454. PMID 20214476
- [Background] Coovadia A, Abrams EJ, Stehlau R, Meyers T, Martens L, Sherman G, Hunt G, Hu CC, Tsai WY, Morris L, Kuhn L. Reuse of nevirapine in exposed HIV-infected children after protease inhibitor-based viral suppression: a randomized controlled trial. JAMA. 2010 Sep 8;304(10):1082-90. doi: 10.1001/jama.2010.1278. PMID 20823434
- [Background] Saez-Llorens X, Violari A, Deetz CO, Rode RA, Gomez P, Handelsman E, Pelton S, Ramilo O, Cahn P, Chadwick E, Allen U, Arpadi S, Castrejon MM, Heuser RS, Kempf DJ, Bertz RJ, Hsu AF, Bernstein B, Renz CL, Sun E. Forty-eight-week evaluation of lopinavir/ritonavir, a new protease inhibitor, in human immunodeficiency virus-infected children. Pediatr Infect Dis J. 2003 Mar;22(3):216-24. doi: 10.1097/01.inf.0000055061.97567.34. PMID 12634581
- [Background] Verweel G, Burger DM, Sheehan NL, Bergshoeff AS, Warris A, van der Knaap LC, Driessen G, de Groot R, Hartwig NG. Plasma concentrations of the HIV-protease inhibitor lopinavir are suboptimal in children aged 2 years and below. Antivir Ther. 2007;12(4):453-8. PMID 17668553
- [Background] Chadwick EG, Capparelli EV, Yogev R, Pinto JA, Robbins B, Rodman JH, Chen J, Palumbo P, Serchuck L, Smith E, Hughes M; P1030 team. Pharmacokinetics, safety and efficacy of lopinavir/ritonavir in infants less than 6 months of age: 24 week results. AIDS. 2008 Jan 11;22(2):249-55. doi: 10.1097/QAD.0b013e3282f2be1d. PMID 18097227
- [Background] Chadwick EG, Pinto J, Yogev R, Alvero CG, Hughes MD, Palumbo P, Robbins B, Hazra R, Serchuck L, Heckman BE, Purdue L, Browning R, Luzuriaga K, Rodman J, Capparelli E; International Maternal Pediatric Adolescent Clinical Trials Group (IMPAACT) P1030 Team. Early initiation of lopinavir/ritonavir in infants less than 6 weeks of age: pharmacokinetics and 24-week safety and efficacy. Pediatr Infect Dis J. 2009 Mar;28(3):215-9. doi: 10.1097/INF.0b013e31818cc053. PMID 19209098
- [Background] Rakhmanina N, van den Anker J, Baghdassarian A, Soldin S, Williams K, Neely MN. Population pharmacokinetics of lopinavir predict suboptimal therapeutic concentrations in treatment-experienced human immunodeficiency virus-infected children. Antimicrob Agents Chemother. 2009 Jun;53(6):2532-8. doi: 10.1128/AAC.01374-08. Epub 2009 Mar 2. PMID 19258274
- [Background] Elsherbiny D, Ren Y, McIlleron H, Maartens G, Simonsson US. Population pharmacokinetics of lopinavir in combination with rifampicin-based antitubercular treatment in HIV-infected South African children. Eur J Clin Pharmacol. 2010 Oct;66(10):1017-23. doi: 10.1007/s00228-010-0847-9. Epub 2010 Jun 16. PMID 20552180
- [Background] Urien S, Firtion G, Anderson ST, Hirt D, Solas C, Peytavin G, Faye A, Thuret I, Leprevost M, Giraud C, Lyall H, Khoo S, Blanche S, Treluyer JM. Lopinavir/ritonavir population pharmacokinetics in neonates and infants. Br J Clin Pharmacol. 2011 Jun;71(6):956-60. doi: 10.1111/j.1365-2125.2011.03926.x. PMID 21564164
- [Background] Palumbo P, Lindsey JC, Hughes MD, Cotton MF, Bobat R, Meyers T, Bwakura-Dangarembizi M, Chi BH, Musoke P, Kamthunzi P, Schimana W, Purdue L, Eshleman SH, Abrams EJ, Millar L, Petzold E, Mofenson LM, Jean-Philippe P, Violari A. Antiretroviral treatment for children with peripartum nevirapine exposure. N Engl J Med. 2010 Oct 14;363(16):1510-20. doi: 10.1056/NEJMoa1000931. PMID 20942667
- [Background] Moorthy A, Kuhn L, Coovadia A, Meyers T, Strehlau R, Sherman G, Tsai WY, Chen YH, Abrams EJ, Persaud D. Induction therapy with protease-inhibitors modifies the effect of nevirapine resistance on virologic response to nevirapine-based HAART in children. Clin Infect Dis. 2011 Feb 15;52(4):514-21. doi: 10.1093/cid/ciq161. Epub 2011 Jan 22. PMID 21258105
- [Background] Eley BS, Meyers T. Antiretroviral therapy for children in resource-limited settings: current regimens and the role of newer agents. Paediatr Drugs. 2011 Oct 1;13(5):303-16. doi: 10.2165/11593330-000000000-00000. PMID 21888444
- [Background] McIlleron H, Willemse M, Werely CJ, Hussey GD, Schaaf HS, Smith PJ, Donald PR. Isoniazid plasma concentrations in a cohort of South African children with tuberculosis: implications for international pediatric dosing guidelines. Clin Infect Dis. 2009 Jun 1;48(11):1547-53. doi: 10.1086/598192. PMID 19392636
- [Background] Schaaf HS, Willemse M, Cilliers K, Labadarios D, Maritz JS, Hussey GD, McIlleron H, Smith P, Donald PR. Rifampin pharmacokinetics in children, with and without human immunodeficiency virus infection, hospitalized for the management of severe forms of tuberculosis. BMC Med. 2009 Apr 22;7:19. doi: 10.1186/1741-7015-7-19. PMID 19386087
- [Background] Thee S, Detjen A, Wahn U, Magdorf K. Pyrazinamide serum levels in childhood tuberculosis. Int J Tuberc Lung Dis. 2008 Sep;12(9):1099-101. PMID 18713511
- [Background] Donald PR, Maher D, Maritz JS, Qazi S. Ethambutol dosage for the treatment of children: literature review and recommendations. Int J Tuberc Lung Dis. 2006 Dec;10(12):1318-30. PMID 17167947
- [Background] Thee S, Seddon JA, Donald PR, Seifart HI, Werely CJ, Hesseling AC, Rosenkranz B, Roll S, Magdorf K, Schaaf HS. Pharmacokinetics of isoniazid, rifampin, and pyrazinamide in children younger than two years of age with tuberculosis: evidence for implementation of revised World Health Organization recommendations. Antimicrob Agents Chemother. 2011 Dec;55(12):5560-7. doi: 10.1128/AAC.05429-11. Epub 2011 Oct 3. PMID 21968358
- [Background] Berenguer J, Perez-Elias MJ, Bellon JM, Knobel H, Rivas-Gonzalez P, Gatell JM, Miguelez M, Hernandez-Quero J, Flores J, Soriano V, Santos I, Podzamczer D, Sala M, Camba M, Resino S; Spanish Abacavir, Lamivudine, and Zidovudine Cohort Study Group. Effectiveness and safety of abacavir, lamivudine, and zidovudine in antiretroviral therapy-naive HIV-infected patients: results from a large multicenter observational cohort. J Acquir Immune Defic Syndr. 2006 Feb 1;41(2):154-9. doi: 10.1097/01.qai.0000194231.08207.8a. PMID 16394846
- [Background] Shey M, Kongnyuy EJ, Shang J, Wiysonge CS. A combination drug of abacavir-lamivudine-zidovudine (Trizivir) for treating HIV infection and AIDS. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD005481. doi: 10.1002/14651858.CD005481.pub2. PMID 19588374
- [Background] la Porte CJ, Colbers EP, Bertz R, Voncken DS, Wikstrom K, Boeree MJ, Koopmans PP, Hekster YA, Burger DM. Pharmacokinetics of adjusted-dose lopinavir-ritonavir combined with rifampin in healthy volunteers. Antimicrob Agents Chemother. 2004 May;48(5):1553-60. doi: 10.1128/AAC.48.5.1553-1560.2004. PMID 15105105
- [Background] Decloedt EH, McIlleron H, Smith P, Merry C, Orrell C, Maartens G. Pharmacokinetics of lopinavir in HIV-infected adults receiving rifampin with adjusted doses of lopinavir-ritonavir tablets. Antimicrob Agents Chemother. 2011 Jul;55(7):3195-200. doi: 10.1128/AAC.01598-10. Epub 2011 May 2. PMID 21537021
- [Background] Ren Y, Nuttall JJ, Egbers C, Eley BS, Meyers TM, Smith PJ, Maartens G, McIlleron HM. Effect of rifampicin on lopinavir pharmacokinetics in HIV-infected children with tuberculosis. J Acquir Immune Defic Syndr. 2008 Apr 15;47(5):566-9. doi: 10.1097/QAI.0b013e3181642257. PMID 18197120
- [Background] Frohoff C, Moodley M, Fairlie L, Coovadia A, Moultrie H, Kuhn L, Meyers T. Antiretroviral therapy outcomes in HIV-infected children after adjusting protease inhibitor dosing during tuberculosis treatment. PLoS One. 2011 Feb 23;6(2):e17273. doi: 10.1371/journal.pone.0017273. PMID 21383838
- [Background] Rae JM, Johnson MD, Lippman ME, Flockhart DA. Rifampin is a selective, pleiotropic inducer of drug metabolism genes in human hepatocytes: studies with cDNA and oligonucleotide expression arrays. J Pharmacol Exp Ther. 2001 Dec;299(3):849-57. PMID 11714868
- [Background] Zhang C, McIlleron H, Ren Y, van der Walt JS, Karlsson MO, Simonsson US, Denti P. Population pharmacokinetics of lopinavir and ritonavir in combination with rifampicin-based antitubercular treatment in HIV-infected children. Antivir Ther. 2012;17(1):25-33. doi: 10.3851/IMP1915. PMID 22267466
- [Background] Anderson BJ, Holford NH. Mechanism-based concepts of size and maturity in pharmacokinetics. Annu Rev Pharmacol Toxicol. 2008;48:303-32. doi: 10.1146/annurev.pharmtox.48.113006.094708. PMID 17914927
- [Background] Holford N. Dosing in children. Clin Pharmacol Ther. 2010 Mar;87(3):367-70. doi: 10.1038/clpt.2009.262. Epub 2010 Jan 20. No abstract available. PMID 20090674
- [Background] Price PS, Conolly RB, Chaisson CF, Gross EA, Young JS, Mathis ET, Tedder DR. Modeling interindividual variation in physiological factors used in PBPK models of humans. Crit Rev Toxicol. 2003;33(5):469-503. PMID 14594104
- [Background] Zar HJ, Cotton MF, Strauss S, Karpakis J, Hussey G, Schaaf HS, Rabie H, Lombard CJ. Effect of isoniazid prophylaxis on mortality and incidence of tuberculosis in children with HIV: randomised controlled trial. BMJ. 2007 Jan 20;334(7585):136. doi: 10.1136/bmj.39000.486400.55. Epub 2006 Nov 3. PMID 17085459
- [Background] Hartkoorn RC, Kwan WS, Shallcross V, Chaikan A, Liptrott N, Egan D, Sora ES, James CE, Gibbons S, Bray PG, Back DJ, Khoo SH, Owen A. HIV protease inhibitors are substrates for OATP1A2, OATP1B1 and OATP1B3 and lopinavir plasma concentrations are influenced by SLCO1B1 polymorphisms. Pharmacogenet Genomics. 2010 Feb;20(2):112-20. doi: 10.1097/FPC.0b013e328335b02d. PMID 20051929
- [Background] Chigutsa E, Visser ME, Swart EC, Denti P, Pushpakom S, Egan D, Holford NH, Smith PJ, Maartens G, Owen A, McIlleron H. The SLCO1B1 rs4149032 polymorphism is highly prevalent in South Africans and is associated with reduced rifampin concentrations: dosing implications. Antimicrob Agents Chemother. 2011 Sep;55(9):4122-7. doi: 10.1128/AAC.01833-10. Epub 2011 Jun 27. PMID 21709081
- [Background] Svard J, Spiers JP, Mulcahy F, Hennessy M. Nuclear receptor-mediated induction of CYP450 by antiretrovirals: functional consequences of NR1I2 (PXR) polymorphisms and differential prevalence in whites and sub-Saharan Africans. J Acquir Immune Defic Syndr. 2010 Dec 15;55(5):536-49. doi: 10.1097/QAI.0b013e3181f52f0c. PMID 20861742
- [Background] Shimizu M, Fukami T, Kobayashi Y, Takamiya M, Aoki Y, Nakajima M, Yokoi T. A novel polymorphic allele of human arylacetamide deacetylase leads to decreased enzyme activity. Drug Metab Dispos. 2012 Jun;40(6):1183-90. doi: 10.1124/dmd.112.044883. Epub 2012 Mar 13. PMID 22415931
- [Background] Nakajima A, Fukami T, Kobayashi Y, Watanabe A, Nakajima M, Yokoi T. Human arylacetamide deacetylase is responsible for deacetylation of rifamycins: rifampicin, rifabutin, and rifapentine. Biochem Pharmacol. 2011 Dec 1;82(11):1747-56. doi: 10.1016/j.bcp.2011.08.003. Epub 2011 Aug 12. PMID 21856291
- [Background] Wiseman CA, Gie RP, Starke JR, Schaaf HS, Donald PR, Cotton MF, Hesseling AC. A proposed comprehensive classification of tuberculosis disease severity in children. Pediatr Infect Dis J. 2012 Apr;31(4):347-52. doi: 10.1097/INF.0b013e318243e27b. PMID 22315002
- [Background] Nijland HM, L'homme RF, Rongen GA, van Uden P, van Crevel R, Boeree MJ, Aarnoutse RE, Koopmans PP, Burger DM. High incidence of adverse events in healthy volunteers receiving rifampicin and adjusted doses of lopinavir/ritonavir tablets. AIDS. 2008 May 11;22(8):931-5. doi: 10.1097/QAD.0b013e3282faa71e. PMID 18453852
- [Background] Dansirikul C, Silber HE, Karlsson MO. Approaches to handling pharmacodynamic baseline responses. J Pharmacokinet Pharmacodyn. 2008 Jun;35(3):269-83. doi: 10.1007/s10928-008-9088-2. Epub 2008 Apr 30. PMID 18446428
- [Background] Gupta P, Hutmacher MM, Frame B, Miller R. An alternative method for population pharmacokinetic data analysis under noncompliance. J Pharmacokinet Pharmacodyn. 2008 Apr;35(2):219-33. doi: 10.1007/s10928-008-9085-5. Epub 2008 Feb 26. PMID 18299967
- [Background] Zhang C, Denti P, Decloedt EH, Ren Y, Karlsson MO, McIlleron H. Model-based evaluation of the pharmacokinetic differences between adults and children for lopinavir and ritonavir in combination with rifampicin. Br J Clin Pharmacol. 2013 Nov;76(5):741-51. doi: 10.1111/bcp.12101. PMID 23432610
- [Derived] Galileya LT, Wasmann RE, Chabala C, Rabie H, Lee J, Njahira Mukui I, Hesseling A, Zar H, Aarnoutse R, Turkova A, Gibb D, Cotton MF, McIlleron H, Denti P. Evaluating pediatric tuberculosis dosing guidelines: A model-based individual data pooled analysis. PLoS Med. 2023 Nov 21;20(11):e1004303. doi: 10.1371/journal.pmed.1004303. eCollection 2023 Nov. PMID 37988391
- [Derived] Rabie H, Tikiso T, Lee J, Fairlie L, Strehlau R, Bobat R, Liberty A, McIlleron H, Andrieux-Meyer I, Cotton M, Lallemant M, Denti P. Abacavir Exposure in Children Cotreated for Tuberculosis with Rifampin and Superboosted Lopinavir-Ritonavir. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e01923-19. doi: 10.1128/AAC.01923-19. Print 2020 Apr 21. PMID 32071055
- [Derived] Rabie H, Denti P, Lee J, Masango M, Coovadia A, Pillay S, Liberty A, Simon F, McIlleron H, Cotton MF, Lallemant M. Lopinavir-ritonavir super-boosting in young HIV-infected children on rifampicin-based tuberculosis therapy compared with lopinavir-ritonavir without rifampicin: a pharmacokinetic modelling and clinical study. Lancet HIV. 2018 Dec 6:S2352-3018(18)30293-5. doi: 10.1016/S2352-3018(18)30293-5. Online ahead of print. PMID 30529029